CLINICAL TRIAL: NCT00215813
Title: An Open-Label Study Of Poly I:Poly C12U (AMPLIGEN®) in Patients With Severely Debilitating Chronic Fatigue Syndrome (CFS)
Brief Title: Ampligen in Chronic Fatigue Syndrome
Status: Temporarily not available | Type: Expanded Access
Sponsor: AIM ImmunoTech Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AMP 511
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Chronic Fatigue Syndrome
Keywords: Chronic Fatigue Syndrome; CFS; ME; Ampligen; poly I:poly C12U; Rintatolimod
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — poly(I).poly(c12,U)

STUDY DESIGN:
Expanded Access Types: Intermediate, Treatment

INTERVENTIONS:
Drug: Poly I: Poly C12U (Rintatolimod) — 200-400 mg IV infusions given twice weekly over a period of 30-60 minutes
  Other Names: Ampligen; Rintatolimod

SUMMARY:
This is an open label study of Ampligen in patients with chronic fatigue syndrome.

DETAILED DESCRIPTION:
An Open-Label Study of Poly I: Poly C12U (Ampligen®) in Patients with Severely Debilitating Chronic Fatigue Syndrome (CFS)/Myalgic Encephalomyelitis (ME). The FDA approved the study for cost recovery. Patients enrolled in the study are responsible for costs related to the therapy, e.g., drug cost, infusion cost, cost of supplies, diagnostic and other laboratory testing.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Chronic Fatigue Syndrome (>= 12 months) as defined by the 1988 Centers for Disease Control and Prevention CDC case definition for CFS or as defined only by the 1994 CDC case definition of CFS (Fukuda et al., Ann Intern Med. 1994; 121:953-959) (other clinical conditions which could present with similar symptoms must be excluded.).
2. Age Range: >= 18 years old, <= 70 years old.
3. Males or non-pregnant, non-lactating females: Females must be of non-child bearing potential (either post-menopausal for two years or surgically sterile including tubal ligation) or using an effective means of contraception (birth control pills, intrauterine device, diaphragm). Alternatively, female patients with a male partner having a successful vasectomy (considered successful if a volunteer reports that a male partner has either documentation of azoospermia by microscopy or a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity post-vasectomy).Females who are less than two (2) years post-menopausal, those with tubal ligations and those using contraception must have a negative serum pregnancy test at baseline within the four (4) weeks prior to the first study medication infusion. Every four weeks, and at study termination a pregnancy test should be performed, either serum or urine stick test. However, if the urine result is positive, a serum pregnancy test will be performed. Females of child bearing potential agree to use an effective means of contraception from four (4) weeks prior to the baseline pregnancy test until four (4) weeks after the last study medication infusion. All male patients agree not to be a sperm donor and to use an effective means of contraception while on study medication and until 90 days after the last study medication infusion.
4. A reduced quality of life as determined by a Karnofsky performance score (KPS) of >= 20 and <= 60. The KPS must be rounded in increments of ten (10).
5. Ability to provide written informed consent indicating awareness of the investigational nature of this study.
6. Documentation (during baseline or historically following the onset of CFS) of a negative ANA or a negative anti-ds (double-stranded) DNA, a negative Rheumatoid Factor, and an erythrocyte sedimentation rate (ESR). Documentation during baseline of a normal T4 (or other laboratory evidence that subject is euthyroid) is also required.
7. Laboratory confirmed negative SARS-CoV-2 (COVID-19) infection by a government approved test / kit within 2 weeks prior to starting study drug dosing.
8. Patients with post-COVID-19 chronic fatigue (PCCF) must meet the 1988 or 1994 CFS CDC Definition for Chronic Fatigue Syndrome except for the duration of the fatiguing illness which must have continued for at least 3 months and must not have preceded the onset of the COVID-19 symptoms. The patient must also have at least one of the following "Long Hauler" symptoms which must have persisted or recurred during 3 or more consecutive months of illness and must not have preceded the onset of the COVID-19 symptoms (fever or chills, cough, shortness of breath or difficulty breathing, new loss of taste or smell or chest pain). Since many patients with mild or no COVID-19 symptoms were not tested for the presence of SARS-CoV-2, many patients with post-COVID-19 chronic fatigue (PCCF) also called "Long Haulers", will not have a history of a positive SARS-CoV-2 test result. A positive serum antibody test for SARS-CoV-2 will be sufficient in these cases.

Exclusion Criteria:

1. Inability to return for scheduled treatment and assessments.
2. Chronic or intercurrent acute medical disorder or disease making implementation or interpretation of the protocol or results difficult or unsafe.
3. Pregnant or lactating females.
4. Therapy with interferons, interleukins, or other cytokines or investigational drugs within 6 weeks of beginning study medication. Subjects must give written informed consent prior to discontinuation of investigational drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Peterson, M.D., Principal Investigator — Sierra Internal Medicine; Vincent F. Hillman, M.D., Principal Investigator — Hunter-Hopkins Center, P.A.
Locations (2):
- United States (2):
  - Sierra Internal Medicine, Incline Village, Nevada
  - Hunter-Hopkins Center, PA, Charlotte, North Carolina

REFERENCES:
- [Background] Strayer DR, Carter WA, Stouch BC, Stevens SR, Bateman L, Cimoch PJ, Lapp CW, Peterson DL; Chronic Fatigue Syndrome AMP-516 Study Group; Mitchell WM. A double-blind, placebo-controlled, randomized, clinical trial of the TLR-3 agonist rintatolimod in severe cases of chronic fatigue syndrome. PLoS One. 2012;7(3):e31334. doi: 10.1371/journal.pone.0031334. Epub 2012 Mar 14. PMID 22431963
- [Background] Strayer DR, Young D, Mitchell WM. Effect of disease duration in a randomized Phase III trial of rintatolimod, an immune modulator for Myalgic Encephalomyelitis/Chronic Fatigue Syndrome. PLoS One. 2020 Oct 29;15(10):e0240403. doi: 10.1371/journal.pone.0240403. eCollection 2020. PMID 33119613
- See also: research — http://www.aimimmuno.com